CLINICAL TRIAL: NCT05900167
Title: Feeding Intolerance Risk Prediction Model in Patients With Enteral Nutrition Through Nasogastric Tube
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiao Jie Chen (Other)
Responsible Party: Sponsor-Investigator, Xiao Jie Chen, Nurse, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: IIT-2023-0054
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Enteral Nutrition
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- enteral nutrition group
  Interventions: Behavioral: enteral nutrition

INTERVENTIONS:
Behavioral: enteral nutrition — The nutritional status of the patient is assessed by the physician to determine the need for enteral nutrition

SUMMARY:
To explore the risk factors of enteral feeding intolerance in critically ill patients, build a risk prediction model and verify it, in order to provide reference for early identification and screening of high-risk groups

DETAILED DESCRIPTION:
Based on the previous literature study, the risk factors of enteral feeding intolerance in critically ill patients were obtained, and the general demographic, disease and treatment information of patients were collected. Four machine learning algorithms, namely traditional logistic regression, random forest, support vector machine and naive Bayes, were used to construct risk prediction models, and the optimal model was selected and verified by comparing the model performance

ELIGIBILITY:
Inclusion Criteria:

* The nutritional status of the patient is assessed by the doctor and the need for enteral nutrition is determined;Patients with first nasogastric tube insertion and successful enteral feeding;There was no gastrointestinal discomfort before enteral nutrition;Patients (or family members) authorized to participate in this study and signed informed consent

Exclusion Criteria:

* Previous gastrointestinal disease or gastrointestinal surgery;enteral nutrition through gastrostomy tube or jejunostomy tube;discontinuation or suspension of enteral nutrition for special reasons other than feeding intolerance;Patients with serious lack of clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size calculation method of this study was based on the results of previous literature studies to obtain enteral nutritional feeding intolerance According to the sample size estimation method of N= [(risk variable) ×(5 ~ 10)]
  ,the incidence of feeding intolerance was 41.3%,so at least 269 samples are needed for further examination.Considering a 10% loss of follow-up rate, the estimated sample size is 299 cases, the data collected in this part of the study as the model Develop the data set.Using the ratio of modeling group: test group = 7:3, and considering 10% loss of follow-up rate, the minimum sample of test group was 143 cases. Therefore, a total of at least 442 samples are needed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 442 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Feeding intolerance | Follow-up was considered complete when the patient reached 7 days of enteral nutrition, the patient was transferred from the ICU, or the patient experienced nutritional interruption for other reasons
  Any symptoms of gastrointestinal adverse reactions are defined as feeding intolerance

IPD SHARING:
Plan to Share IPD: No